CLINICAL TRIAL: NCT01993394
Title: Influence of Hyperoxia and Hypergravity on Pulmonary Ventilation and Perfusion
Brief Title: Effect of Hyperoxia and Hypergravity on Lung Ventilation and Perfusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Direction Centrale du Service de Santé des Armées (Other)
Collaborators: Val de Grâce Hospital (Unknown); Uppsala University Hospital (Other)
Responsible Party: Principal Investigator, Stéphanie Montmerle-Borgdorff, researcher, Direction Centrale du Service de Santé des Armées
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: 10co706
Record Dates: First submitted 2013-11-14; First posted 2013-11-25 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Atelectasis
Keywords: human centrifuge, oxygen, imaging, stroke volume, lung
MeSH Terms: conditions — Pulmonary Atelectasis | interventions — Hypergravity; nitrox

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- ventilation (Experimental): hypergravity gas mixture
  Interventions: Other: hypergravity; Other: gas mixture

INTERVENTIONS:
Other: hypergravity — 1hr sitting rest followed by 10 min of hypergravity (2 centrifuge runs)
Other: gas mixture — breathing air, 44.5%O2 or 100%O2

SUMMARY:
The primary aim of this project is to get further knowledge on the effects of + Gz accelerations and hyperoxia on lung ventilation in humans. The secondary aim is to study lung perfusion and cardiovascular function in these conditions.

DETAILED DESCRIPTION:
Experiments were conducted in a human centrifuge. The protocol aimed at mimicking a routine peacetime flight in combat aircraft, and included 10-min exposure to +1.4 - +3.5 Gz. Subjects were exposed three times to this sequence, breathing air, 44.5% O2 or 100% O2.

Ten volunteers wearing anti-G trousers participated in the study. The Ethics Committee Ile-de-France III and the French National Agency for Drug Safety (ANSM) approved the protocol (number 2009-A01092-55).

Three different imaging techniques, electrical impedance tomography (EIT), pulmonary ultrasound and chest SPECT/CT were used and compared. EIT enabled ventilation monitoring in the human centrifuge, whereas pulmonary ultrasound and SPECT/CT gave functional and topographical information before and after exposure to +Gz accelerations. EIT analysis focused on regional ventilation, SPECT on global lung ventilation and perfusion, CT on the presence of atelectasis, and pulmonary ultrasound analysis looked for comet tails in 64 chest areas. Arterial blood pressure was recorded continuously by finger photoplethysmography. Cardiac output and stroke volume were computed from these recordings, using three different algorithms. Echocardiography was used as reference non-invasive technique for stroke volume determination and performed before and after exposure to +Gz accelerations.

ELIGIBILITY:
Inclusion Criteria:

* normal lung function checked by pulmonary function tests

Part 1 exclusion Criteria:

* past medical history of heart or lung disease
* current medical treatment for heart or lung disease
* smoking
* bad tolerance to +Gz accelerations (G-induced loss of consciousness, motion sickness)

Part 2 exclusion criteria:

* past medical history of heart or lung disease
* current medical treatment for heart or lung disease
* smoking
* The use of medication for hypertension
* asymmetric values of left/right humeral arterial blood pressure
* significant echocardiographic abnormalities or bad echogenicity
* bad tolerance to +Gz accelerations (G-induced loss of consciousness, motion sickness)

Ages: 25 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2011-10; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
change in regional ventilation distribution | baseline, 2hrs 30min
  "per lobe and per quadrant at 5th intercostal space level"

SECONDARY OUTCOMES:
change in regional pulmonary perfusion | baseline, 2hrs 30min
  "per lobe and per quadrant at 5th intercostal space level"
cardiac output (L/min) | 2hrs
  "echocardiography (sub-aortic diameter), photoplethysmography (Liljestrand, systolic area and Windkessel algorithms)"

OTHER OUTCOMES:
tidal volume | 2hrs 30min
  global (mL, area under the flow versus time curve) and regional (% change per quadrant at 5th intercostal space level)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Garin, MD, PhD, Study Chair — Armed Forces Biomedical Research Institute
Locations (2):
- France (2):
  - Armed Forces Biomedical Research Institute, Brétigny-sur-Orge
  - Department of Nuclear Medicine, Val-de-Grâce hospital, Paris